CLINICAL TRIAL: NCT06010940
Title: Impact of Physical Therapy of Dysphagia on Preventing Pneumonia in Acute Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, heba ahmed khalifa, Ass. Prof. Dr of Physical therapy for Neurology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/002939
Record Dates: First submitted 2023-08-17; First posted 2023-08-25 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Stroke, Acute; Dysphagia; Pneumonia
MeSH Terms: conditions — Stroke; Deglutition Disorders; Pneumonia | interventions — Dietary Supplements; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): Control group (A) was treated by nasogastric tube and oral care.
  Interventions: Dietary Supplement: Dietary supplement
- study group (Experimental): Study group (B) was treated as the control group in addition to a designed physical therapy program consisting of neuromuscular electrical stimulation in addition to exercises for oropharyngeal muscles.
  Interventions: Dietary Supplement: Dietary supplement; Other: Physical therapy

INTERVENTIONS:
Dietary Supplement: Dietary supplement — nasogastric tube and oral care
Other: Physical therapy — Designed physical therapy program consisting of neuromuscular electrical stimulation in addition to exercises for oropharyngeal muscles.
  Arms: study group

SUMMARY:
To investigate the impact of physical therapy intervention of dysphagia on preventing pneumonia in acute stroke patients

DETAILED DESCRIPTION:
Seventy acute ischemic cerebrovascular stroke patients suffering from dysphagia were selected from the stroke unit in El-Kasr EL Ainy Hospital. Their ages ranged from 49 -65 years. Stroke dysphagia was diagnosed by a neurologist. Gugging swallowing screen and A2DS2 score was used to assess risk of developing pneumonia. Stroke associated pneumonia was diagnosed by: Recommended Diagnostic Criteria for Definite and Probable SAP in Patients Not Receiving Mechanical Ventilation Based on the CDC Criteria. The selected patients were randomly assigned into two equal groups control group (A) and study group (B). Control group (A) was treated by nasogastric tube and oral care. Study group (B) was treated as the control group in addition to a designed physical therapy program consisting of neuromuscular electrical stimulation in addition to exercises for oropharyngeal muscles. Assessment was done before treatment, at the middle and at the end of treatment for each patient. Treatment was conducted for five sessions per week for one month.

ELIGIBILITY:
Inclusion Criteria:

* All patients were diagnosed of stroke dysphagia by a neurologist.
* Severity of stroke ranged from mild to moderate according to NIHSS score (NIHSS less than or equal 16).
* Patients' age ranged from 49 to 65 years old.
* Patients had the ability to understand and follow instructions.
* Patients were able to sit in upright position.

Exclusion Criteria:

* History of previous stroke.
* History of any swallowing problem.
* History of any disease, head and neck surgery or tumor that causes swallowing dysfunction.
* Any lung disease or pneumonia on admission.
* Patients with cognitive deficits or disturbed conscious level.
* Patients on mechanical ventilator.
* Patients with sensory or global aphasia.

Ages: 49 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-10-11 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
The Gugging swallowing screen test score | at baseline
  Test used to detect dysphagia and aspiration risk. Score ranged from 0 to 20 where 0 indicates sever dysphagia and 20 indicates normal swallowing
The Gugging swallowing screen test score | At middle of intervention (after two weeks)
  Test used to detect dysphagia and aspiration risk. Score ranged from 0 to 20 where 0 indicates sever dysphagia and 20 indicates normal swallowing
The Gugging swallowing screen test score | post intervention (after one month)
  est used to detect dysphagia and aspiration risk. Score ranged from 0 to 20 where 0 indicates sever dysphagia and 20 indicates normal swallowing

SECONDARY OUTCOMES:
Incidence of participant with stroke associated pneumonia | at baseline
  Measuring number and percentage of participants with stroke associated pneumonia in each group
Incidence of participant with stroke associated pneumonia | At middle of intervention (after two weeks)
  Measuring number and percentage of participants with stroke associated pneumonia in each group
Incidence of participant with stroke associated pneumonia | post intervention (after one month)
  Measuring number and percentage of participants with stroke associated pneumonia in each group

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dziewas R, Michou E, Trapl-Grundschober M, Lal A, Arsava EM, Bath PM, Clave P, Glahn J, Hamdy S, Pownall S, Schindler A, Walshe M, Wirth R, Wright D, Verin E. European Stroke Organisation and European Society for Swallowing Disorders guideline for the diagnosis and treatment of post-stroke dysphagia. Eur Stroke J. 2021 Sep;6(3):LXXXIX-CXV. doi: 10.1177/23969873211039721. Epub 2021 Oct 13. PMID 34746431
- [Background] Lo YK, Fu TC, Chen CP, Yuan SS, Hsu CC. Involvement of swallowing therapy is associated with improved long-term survival in patients with post-stroke dysphagia. Eur J Phys Rehabil Med. 2019 Dec;55(6):728-734. doi: 10.23736/S1973-9087.19.05893-3. PMID 31958220